CLINICAL TRIAL: NCT00455949
Title: Effect of Premature Luteinization on the Oocyte Quality in Oocyte Donation Program.
Status: Completed | Type: Observational
Sponsor: Instituto Valenciano de Infertilidad, IVI VALENCIA (Other)
Other Study IDs: VLC-MM-0106-307-14
Record Dates: First submitted 2007-04-03; First posted 2007-04-04 (Estimated); Last update posted 2007-04-04 (Estimated); Status verified 2007-04

CONDITIONS: Premature Luteinization

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Analyze the possible effect of the progesterone levels of the hCG administration on the oocyte embryo quality. The primary endpoint of this study is the pregnancy rate.

ELIGIBILITY:
Inclusion Criteria:

* Oocyte donors; age range: 18 - 34; BMI: 18 - 29; long protocol.

Exclusion Criteria:

* PCO syndrome;

Ages: 18 Years to 34 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult

CONTACTS AND LOCATIONS:
Overall Officials: Marco Melo, MD, Principal Investigator — Instituto Valenciano de Infertilidad
Locations (1):
- Instituto Valenciano de la Infertilidad, Valencia, Valencia, Spain